CLINICAL TRIAL: NCT04823819
Title: Assessment of Effectiveness and Safety of Transcranial Magnetic Stimulation (rTMS) Combined With Transcranial Direct Current Stimulation (tDCS) in Dementia Treatment in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Jakub Kazmierski, PhD, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNN/246/20/KE
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rTMS stimulation (Active Comparator): 20 sessions of stimulation with increasing intensity, reaching maximum in the 4th session.
  Interventions: Device: Magnetic Stimulator DuoMag
- tDCS stimulation (Active Comparator): The stimulation time will be 20 minutes, the current intensity will be 2mA.
  Interventions: Device: neuroConn DC-STIMULATOR
- Sham rTMS stimulation (Sham Comparator): 20 sessions of stimulation, but without current.
  Interventions: Device: Magnetic Stimulator DuoMag
- Sham tDCS stimulation (Sham Comparator): The stimulation time will be 20 minutes, but without current.
  Interventions: Device: neuroConn DC-STIMULATOR

INTERVENTIONS:
Device: Magnetic Stimulator DuoMag — Stimulation of the left dorsolateral prefrontal cortex
  Arms: Sham rTMS stimulation; rTMS stimulation
Device: neuroConn DC-STIMULATOR — One electrode (anode) will be placed on the left dorsolateral prefrontal cortex, the other (cathode) on the right temporal lobe.
  Arms: Sham tDCS stimulation; tDCS stimulation

SUMMARY:
Alzheimer's disease is the most common disease responsible for dementia, accounting for 40-70% of all dementia cases. Alzheimer's disease is characterized by a gradual and slow decline in memory and other cognitive functions and activities.

The medications currently used in Alzheimer's disease were introduced in the 1990s and exhibit insufficient effectiveness. Despite their use, the disease rapidly progresses, leading to complete loss of independence and death. There are conducted numerous studies on new molecules, however none of them has been successfully accomplished so far. Transcranial magnetic stimulation (TMS) is one of the youngest electrophysiological methods, enabling non-invasive and painless stimulation of the central and peripheral nervous system. Another non-invasible neurophysiological method that is utilized in treating patients with neurological dysfunctions and mental disorders is Transcranial direct current stimulation (tDCS). Clinical trials conducted with isolated usage of rTMS and tDCS showed a positive effect of these methods on the enhancement of cognitive functions in patients with Alzheimer's disease.

The aim of the project is to evaluate the effectiveness and safety of the combination of Repetitive Transcranial Magnetic Resonance (rTMS) with Transcranial direct current stimulation in the treatment of Alzheimer's dementia. The primary goal of the project is to assess whether the use of combined tDCS and rTMS therapies in patients diagnosed with mild to moderate Alzheimer's disease improves patients' cognitive functions, including memory, attention, thinking, executive and language functions. The research hypothesis assumes that the combination of rTMS and tDCS therapy is an effective method of Alzheimer's disease therapy that can improve cognitive functions and functioning of patients, both in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate dementia in Alzheimer's disease, diagnosed using DSM-5 criteria.
* MMSE score from 12 to 26 points
* ADAS-Cog over 17 points
* Voluntary consent to participate in the study
* there is a related person or legal guardian who consented to assist the patient in the course of the study
* Minimum 8 years of education.
* It is allowed to use cholinesterase inhibitors and / or memantine for at least 3 months prior to study entry and at a stable dose for at least 60 days prior to study entry.

Exclusion Criteria:

* Severe agitation
* Intellectual Disability
* Informed consent is not possible
* Unstable somatic condition
* Use of benzodiazepines or barbiturates 2 weeks prior to screening
* Participation in a clinical trial with coinciding factors within 6 months prior to the start of the trial
* Seizures
* Contraindications to rTMS treatment according to the rTMS questionnaire attached to the protocol
* Contraindications to tDCS treatment according to the tDCS questionnaire attached to the protocol
* Patients with depression, bipolar, or psychotic disorders, or any other neurological or psychiatric condition (current or past) that the Investigator considers to be interfering with the study
* Alcoholism or drug addiction as defined by DSM-5 in the last 5 years (addicted for more than a year and or in remission for less than 3 years)
* Patients with any medical condition that the Investigator considers to be an exclusion criterion from the study

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
MMSE Scale | up to 12 weeks
  Assessment conducted on baseline, up to 1 week after end of the procedure and after 12 weeks.
ADAS-Cog Scale | up to 12 weeks
  Assessment conducted on baseline, up to 1 week after end of the procedure and after 12 weeks.
NPI Scale | up to 12 weeks
  Assessment conducted on baseline, up to 1 week after end of the procedure and after 12 weeks.
ADCS | up to 12 weeks
  Assessment conducted on baseline, up to 1 week after end of the procedure and after 12 weeks.
GDS | up to 12 weeks
  Assessment conducted on baseline, up to 1 week after end of the procedure and after 12 weeks.
Zarit Burden Interview | up to 12 weeks
  Assessment conducted on baseline, up to 1 week after end of the procedure and after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Kazmierski, PhD, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Department of Old Age Psychiatry and Psychotic Disorders Medical University of Lodz, Lodz, Poland